CLINICAL TRIAL: NCT06391476
Title: Morbi-mortality and Development at 2 Years in Infants Born at the Limit of Viability
Brief Title: Prematurity at the Limit of Viability
Acronym: PRELIVIA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2024_001
Record Dates: First submitted 2024-04-04; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Very Preterm Maturity of Infant
Keywords: Prematurity; Morbi-mortality; Neurosensory development
MeSH Terms: conditions — Premature Birth | interventions — Gestational Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extremely preterm infants, born between 22 and 25 weeks gestational age: Infant born between 22 and 25 weeks gestational age and hospitalized at the Croix-Rousse Hospital
  Interventions: Other: Study of the evolution of a cohort of children born between 22 and 25 weeks gestational age

INTERVENTIONS:
Other: Study of the evolution of a cohort of children born between 22 and 25 weeks gestational age — * Study of mortality in a cohort of children born between 22 and 25 weeks gestational age
  * Study of neonatal morbidity
  * Description of postnatal growth
  * Description of nutrition and breastfeeding at discharge
  * Study of the neurological, respiratory and growth outcome at 2 years.

SUMMARY:
Advancements in perinatal care have significantly improved the survival of extremely premature infants, establishing a viability threshold below 25 weeks' gestational age (GA). However, management at the limit of viability poses ethical and decision-making problems for health-care professionals. They grapple with the delicate balance between potential survival and long-term disabilities.

These decisions, as well as the information given to families, are based on knowledge of the prognosis as assessed by national and international epidemiological studies. Healthcare professionals rely on population-based estimations but face discrepancies in predicting outcomes because there are significant variation depending on perinatal center and country where infants are hospitalized. In the large French epidemiological study, 9,6% of livebirths included were born at 22-25 wks and only 38% survived.

In the neonatology department of the croix rousse, these infants have been actively cared for for many years, which has allowed the development of specific skills that are essential for the proper management of these very high-risk patients. Furthermore, EPIPAGE 2 included data from centers where perinatal management was probably not very active at these extreme ages. It results in worse neonatal outcomes as evaluated at the national level than outcomes data evaluated at the neonatal intensive care unit of Croix-Rousse hospital. Using data from EPIPAGE 2 study for clinical decision could lead to avoid active care at the for some infants at the limit of viability It is needed to obtain complete evaluation of neonatal outcomes of infants hospitalized at the Croix-Rousse hospital, so that clinicians may rely on actualized data related to the practices in their perinatal center. It is also needed to compare outcomes with data from large national and international cohorts, to identify and quantify differences. Data about later neurodevelopment outcomes, at 2 years, are also needed as it can taken in consideration in decision-making process.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 22 and 25 weeks gestational age
* Infants hospitalized at the tertiary care neonatal unit of Croix-Rousse hospital
* Infants born between January 2010 and December 2019

Exclusion Criteria:

- None

Ages: 22 Weeks to 25 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely premature newborn (between 22 and 25 weeks gestational age) treated at the Croix-Rousse hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | up to 24 months corrected age
  Proportion of deaths in a cohort of infants born between 22 - 25 weeks gestational age

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Croix Rousse, Lyon, Rhone, France